CLINICAL TRIAL: NCT05079776
Title: Assessing the Use of a Growth Artificial Intelligence Algorithm for Estimating the leNgth of Children in Real-world Setting
Brief Title: Assessing a Length Artificial Intelligence Algorithm to Estimate Length of Children
Acronym: GAIN
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SBB20R&31696
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Growth; Stunting, Nutritional
Keywords: growth; length; artificial intelligence; algorithm
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 0-18 months of age: Children aged 0-18 months of age with no structural abnormalities of the lower limbs or orthopedic conditions
  Interventions: Other: Physical length measurement

INTERVENTIONS:
Other: Physical length measurement — Physical length will be measured and images will be collected for AI to estimate the length

SUMMARY:
An exploratory study to explore the possibility of using computer vision algorithms to estimate a child's length using images taken by a healthcare professional or parents.

DETAILED DESCRIPTION:
This is an exploratory, observational, pilot study that aims to evaluate the performance of a Length Artificial Intelligence (LAI) algorithm in a real world setting. Images will be collected by parents or healthcare professionals, together with physical length measurements. This data will be used to evaluate the accuracy of the algorithm and to explore potential improvements. Data on the acceptance and experience of the using the algorithm will be collected for improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0 to 18 months old.
2. Parent(s) should have access to the internet and a smartphone or tablet to complete study questionnaires, take images and upload images.
3. Parent(s) should be able to comprehend the content of the study and to complete the study questionnaires in English.
4. Written consent from parent.

Exclusion Criteria:

1. Parent(s) incapable of completing the study questionnaires and uploading of the images using smart phone or tablet with internet.
2. Children unable to undergo length measurement (e.g. children with structural abnormalities of the lower limbs or orthopedic conditions such as club foot, hip dysplasia, etc).

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 0-18 months of age with no physical deformities.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of the length AI | 2 days
  Accuracy of the length AI in a clinic and in a home setting, derived from:
  1. The length AI prediction from images collected
  2. The physical length measurement of subjects

SECONDARY OUTCOMES:
Investigator's assessment on collection of images | 2 days
  Investigator's assessment on the ease of collecting the images [Very Easy, Easy, Normal, Difficult, Very Difficult]
Parental acceptability of the length AI | 2 days
  Parental acceptability of length AI assessed via the study questionnaire [Very useful, useful, neutral, not useful, very not useful]
Investigators' (or delegates) acceptability of length AI | 2 days
  Investigators' (or delegates) likelihood of using the length AI assessed via the study questionnaire [Very Likely, Likely, Neutral, Unlikely, Very Unlikely]

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan D, Chua MC, Hadimaja M, Mukherjee S, Wong J, Yap F. Artificial intelligence-driven anthropometric assessment for young children: evaluating the accuracy and practicality of a digital image-based length and weight prediction tool. BMJ Health Care Inform. 2025 Dec 9;32(1):e101540. doi: 10.1136/bmjhci-2025-101540. PMID 41365661
- [Derived] Chua MC, Hadimaja M, Wong J, Mukherjee SS, Foussat A, Chan D, Nandal U, Yap F. Exploring the Use of a Length AI Algorithm to Estimate Children's Length from Smartphone Images in a Real-World Setting: Algorithm Development and Usability Study. JMIR Pediatr Parent. 2024 Nov 22;7:e59564. doi: 10.2196/59564. PMID 39576977